CLINICAL TRIAL: NCT01366911
Title: Can Stem Cells Predict Orthopaedic Outcomes? The Correlation of Bone Density Findings Post Total Hip Arthoplasty With Stem Cell Assays Obtaned at Time of Surgery
Brief Title: Stem Cells Predicting Orthopedic Outcomes
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0168-11-FB
Record Dates: First submitted 2011-05-04; First posted 2011-06-06 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Hip Arthroplasty
Keywords: stem cells; QCT testing; Bone density findings; mesenchymal stem cells

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stem cell & quanitative computed tomography QCT testing: The association between bone mineral denity adjacent to acetabular implants, as measured by quanitative computed tomography (QCT), at least 2 years post Total Hip Arthoplasty (THA) surgery and mesechymal stem cell assays, obtained at time of surgery, will evaluate if stem cells can predict orthopaedic surgical outcomes.
  Detailed Description:
  Subjects who have undergone a THA and who previously consented to "Stem Cell Quality Assays: Correlation with Aging/Health" study which used excess bone marrow and blood samples to complete stem cell assay labs will be invited back at least 2 years post THA to complete bilateral hip x-rays, if not already completed as part of routine medical follow up plus a QCT bone density testing and to complete a questionnaire regarding smoking, alcohol and exercise history along with recording BMIs.

SUMMARY:
This is a pilot study to provide preliminary data of the association between bone mineral denity adjacent to acetabular implants, as measured by quanitative computed tomography (QCT), at least 2 years post Total Hip Arthoplasty (THA) surgery with Mesechymal stem cell assays, obtained at time of surgery, and to begin to evaluate if stem cells can predict orthopaedic surgical outcomes.

DETAILED DESCRIPTION:
Subjects who have undergone a THA and who previously consented to "Stem Cell Quality Assays: Correlation with Aging/Health" study which used excess bone marrow and blood samples to complete stem cell assay labs will be invited back at least 2 years post THA to complete bilateral hip x-rays, if not already completed as part of routine medical follow up plus a QCT bone density testing and to complete a questionnaire regarding smoking, alcohol and exercise history along with recording BMIs.

This ability to identify older individuals with compromised stem cell function could offer opportunities to develop and test new preventative and therapeutic strategies to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* subjects who previously had a total hip arthroplasty and had stem cell assays completed on excess bone marrow

Exclusion Criteria:

* Subjects who do not wish to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Orthopaedic surgical patients at specific clinic
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2011-04-22 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2014-01-10 (Actual)

PRIMARY OUTCOMES:
Can Stem Cells Predict Orthopaedic Outcomes? | Enrollment expected to begin June 2011and this pilot study is expected to be completed by May 2012.
  Bone mineral density adjacent to acetabular implants will be evaluated using QCT which can show early bony changes, which can provide information about the quality of implant fixation and surrounding bone adaption. X-rays will evaluate component loosening, wear, alignmet and osteolytis. Patient characteristics will be summarized using descriptive statistics. Spearman correlation coefficients will be used to assess the association of Mesenchymal stem cell assays and bone density findings.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Garvin, MD, Principal Investigator — UNMC
Locations (1):
- University of Nebraska Medical Center, Orthopaedic Surgery, Omaha, Nebraska, United States